CLINICAL TRIAL: NCT00598897
Title: Open, Noncomparative Trial of Multidrug Regimens Containing Clarithromycin and Rifabutin Administered Three Times Per Week for the Treatment of M. Avium Complex (MAC) Lung Disease
Brief Title: Use of Clarithromycin and Rifabutin for the Treatment of M. Avium Complex (MAC) Lung Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center at Tyler (Other)
Collaborators: Abbott (Industry); Pfizer (Industry)
Responsible Party: Principal Investigator, Richard J. Wallace, Jr., M.D., Chairman Department of Microbiology, The University of Texas Health Science Center at Tyler
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 447
Record Dates: First submitted 2008-01-11; First posted 2008-01-23 (Estimated); Last update posted 2017-05-23 (Actual); Status verified 2017-05

CONDITIONS: Mycobacterium Avium Complex Lung Disease
Keywords: MAC
MeSH Terms: interventions — Clarithromycin; Rifabutin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- clarithromycin and rifabutin/rifampin (Experimental): Clarithromycin and rifabutin/rifampin with ethambutol given three times weekly.
  Interventions: Drug: clarithromycin, rifabutin

INTERVENTIONS:
Drug: clarithromycin, rifabutin — Clarithromycin three times per week (variable dosage) in combination with multiple drugs including rifabutin or rifampin three times per week (variable dosage). Dosage dependent on age, weight and other patient-specific health factors.
  Other Names: Biaxin, mycobutin

SUMMARY:
To determine the safety and tolerance of clarithromycin given three times per week in combination with multiple drugs including rifabutin three times per week

DETAILED DESCRIPTION:
Safety and tolerance of clarithromycin given 3 times weekly with multiple drugs including ethambutol and rifampin/rifabutin

ELIGIBILITY:
Inclusion Criteria:

* Meet American Thoracic Society criteria for nontuberculous mycobacterial lung disease: two or more AFB smear positive, culture positive sputums or bronchoscopic samples and/or two or more AFB smear negative respiratory samples with moderate to heavy growth (2+-4+); abnormal CXR consistent with M. avium lung disease; absence of other potential mycobacterial or fungal lung pathogens (except for the coexistence of M. abscessus).
* Adults age 18 and older
* Pretreatment isolate of M. avium complex available for MIC determination

Exclusion Criteria:

* History of allergy to study drugs
* If a mensruating female, not pregnant and on adequate birth control.
* Children less than 18 years of age
* HIV + or at high risk for HIV infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 1995-08 (Actual); Primary Completion 2002-08-07 (Actual); Study Completion 2017-05-18 (Actual)

PRIMARY OUTCOMES:
Clinical and microbiological outcomes such as clinical symptoms and laboratory cultures | 6 months
  sputum conversion culture neg x3

SECONDARY OUTCOMES:
Clinical and microbiological outcomes | 1 yr
  culture neg 1 yr on treatment

CONTACTS AND LOCATIONS:
Overall Officials: Richard J Wallace Jr., M.D., Principal Investigator — The University of Texas Health Science Center at Tyler
Locations (1):
- The University of Texas Health Science Center at Tyler, Tyler, Texas, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share.